CLINICAL TRIAL: NCT07370350
Title: Standardized Tongue Ultrasound Protocol for Tongue Characteristics in Children and Adolescents With Obesity After a 30-week Inpatient Weight Loss Program
Brief Title: Ultrasound Assessment of Tongue Characteristics in Children and Adolescents With Obesity
Status: Recruiting | Type: Observational
Sponsor: Haute Ecole Bruxelles-Brabant (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Frédéric Paillaugue, Principal Investigator, MSc PT Drs, Haute Ecole Bruxelles-Brabant
Other Study IDs: 93018
Record Dates: First submitted 2026-01-03; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Obesity & Overweight; Pediatric Obesity; Obstructive Sleep Apnea (OSA)
Keywords: Tongue ultrasound; Shear-wave elastography; Pediatric obesity; Obstructive sleep apnea
MeSH Terms: conditions — Obesity; Overweight; Pediatric Obesity; Sleep Apnea, Obstructive | interventions — Body Height; Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Children and adolescents with obesity participating in a specialized inpatient multidisciplinary weight-loss rehabilitation program (30 weeks).
  As this is an observational study, tongue ultrasound (via a submental approach, a non-invasive, risk-free and harmless procedure) will be performed and basic anthropometric data (height, weight, neck circumference, hydration status) will be collected.
  Interventions: Other: Submental ultrasound
- Control group: Healthy children and adolescents. As this is an observational study, tongue ultrasound (via a submental approach, a non-invasive, risk-free and harmless procedure) will be performed and basic anthropometric data (height, weight, neck circumference, hydration status) will be collected.
  Interventions: Other: Submental ultrasound

INTERVENTIONS:
Other: Submental ultrasound — Tongue ultrasound via a submental approach. This non-invasive, risk-free and harmless protocol will study both morphological and dynamic characteristics of the tongue.
  Other Names: Anthropometric measurements (height, weight, neck circumference)

SUMMARY:
This longitudinal observational study aims to validate ultrasound-based tongue markers related to tongue characteristics, including fat accumulation, morphologic and mechanical properties of the tongue in children and adolescents with obesity. Participants are assessed at baseline and after completion of a standardized 30-week inpatient weight-loss rehabilitation program at the Zeepreventorium (De Haan, Belgium). Tongue ultrasound parameters are examined in relation to anthropometric characteristics and obstructive sleep apnea condition.

DETAILED DESCRIPTION:
This prospective observational cohort study investigates ultrasound-based tongue characteristics in children and adolescents with obesity. Participants undergo standardized submental tongue ultrasound examinations at baseline and after completion of a 30-week inpatient multidisciplinary weight-loss rehabilitation program.

Ultrasound measures include tongue morphology, fat-related imaging biomarkers, and mechanical properties assessed using shear-wave elastography. Anthropometric data and validated sleep-disordered breathing questionnaires are collected in parallel. Measurement reliability is evaluated, and associations between ultrasound parameters, anthropometric characteristics, and sleep-related outcomes are explored.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 6 to 18 years
* Diagnosis of obesity
* Already enrolled in the inpatient weight-loss rehabilitation program at the Zeepreventorium
* Written informed consent from legal guardian and assent from the participant, following the legal requirements

Exclusion Criteria:

* Known orthopedic, traumatic, or rheumatologic conditions affecting the cervicocephalic region
* Contraindication to ultrasound examination
* Inability to comply with study procedures
* Inability to understand the procedures

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and adolescents with obesity participating in a specialized inpatient multidisciplinary weight-loss rehabilitation program in Zeepreventorium de Haan.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Tongue stiffness | at baseline and after 30-weeks weight loss program
  Tongue stiffness is measured by shear-wave elastography and expressed in kPa.
Intraclass correlation coefficient, ICC | Baseline
  Intraclass correlation coefficient will be used to assess intra and inter-rater reliability of ultrasound markersUltrasound reliability and repeatability of tongue measurements will be assessed with intraclass correlation coefficients (ICC), along with their 95% confidence intervals. Each ultrasound measurement (tongue size and morphological parameters, echo intensity, stiffness, tissue attenuation imaging, tissue scatter distribution imaging, and fat fraction) in sagittal and coronal planes will be performed twice in fifteen participants by the principal investigator, with a 24-hour interval between examinations.

SECONDARY OUTCOMES:
Tongue thickness | at baseline and after 30 weeks weight loss program
  Tongue thickness (expressed in cm) will be measured with ultrasound as the perpendicular distance from the deep fascia of the geniohyoid muscle to the highest lingual dorsum in the midsagittal plane
Echo Intensity | at baseline and after a 30 weeks weight loss program
  Echo intensity will be measured with ImageJ / Fiji software (ImageJ, US NIH, Bethesda, USA) and refers to the mean value of pixels of an area, based on a grey scale between 0 (black) and 255 (white)
Tissue Attenuation Imaging index | at baseline and after a 30 weeks weight loss program
  Attenuation will be measured with ultrasound and depicts the quantitative measurement of ultrasound attenuation in tissues. It is expressed as an attenuation coefficient in dB/cm/MHz.
OSA-18 questionnaire | Baseline and after a 30-weeks weight loss program
  The Obstructive Sleep Apnea - 18 questionnaire is specific to obstructive sleep apnea in children and will be used for correlation analysis. Quality of life is assessed using the Obstructive Sleep Apnea - 18 Quality of Life Survey (OSA-18), a validated questionnaire comprising 18 items. Total scores range from 18 to 126, with higher scores indicating poorer quality of life and greater disease impact, and lower scores reflecting better outcomes.
Weight | baseline and after a 30 weeks weight loss program
  Weight will be measured with a Tanita scale and expressed in kg
Height | Baseline and after a 30 weeks weight loss program
  Height will be measured with a stadiometer and expressed in cm
BMI Z score | Baseline and after a 30-weeks weight loss program
  BMI Z score will be calculated using combined weight, heigt, sex and age, in reference with CDC tables

CONTACTS AND LOCATIONS:
Overall Officials: Steven Provyn, Prof PhD, Study Director — Haute Ecole Bruxelles Brabant & Vrije Universiteit Brussel
Locations (2):
- Belgium (2):
  - ISEK-HE2B, av. Schalle 91, Brussels
  - Zeepreventorium Koninklijke Baan 5, De Haan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the inclusion of minors and data protection regulations.

REFERENCES:
- [Background] Brockmann, P., & Gozal, D. (2022). Neurocognitive Consequences in Children with Sleep Disordered Breathing: Who Is at Risk? Children, 9(9), 1278. https://doi.org/10.3390/children9091278 Chu, C.-A., Chen, Y.-J., Chang, K.-V., Wu, W.-T., & Özçakar, L. (2021). Reliability of Sonoelastography Measurement of Tongue Muscles and Its Application on Obstructive Sleep Apnea. Frontiers in Physiology, 12, 654667. https://doi.org/10.3389/fphys.2021.654667 da Silva Gusmão Cardoso, T., Pompéia, S., & Miranda, M. C. (2018). Cognitive and behavioral effects of obstructive sleep apnea syndrome in children: A systematic literature review. Sleep Medicine, 46, 46-55. https://doi.org/10.1016/j.sleep.2017.12.020 Gipson, K., Lu, M., & Kinane, T. B. (2019). Sleep-Disordered Breathing in Children. Pediatrics in Review, 40(1), 3-13. https://doi.org/10.1542/pir.2018-0142 Glicksman, A., Hadjiyannakis, S., Barrowman, N., Walker, S., Hoey, L., & Katz, S. L. (2017). Body Fat Distribution Ratios and Obstructive Sleep Apnea Severity in Youth With Obesity. Journal of Clinical Sleep Medicine: JCSM: Official Publication of the American Academy of Sleep Medicine, 13(4), 545-550. https://doi.org/10.5664/jcsm.6538 Halbower, A. C., Degaonkar, M., Barker, P. B., Earley, C. J., Marcus, C. L., Smith, P. L., Prahme, M. C., & Mahone, E. M. (2006). Childhood Obstructive Sleep Apnea Associates with Neuropsychological Deficits and Neuronal Brain Injury. PLoS Medicine, 3(8), e301. https://doi.org/10.1371/journal.pmed.0030301 Yu, J. L., Wiemken, A., Schultz, S. M., Keenan, B. T., Sehgal, C. M., & Schwab, R. J. (2022). A comparison of ultrasound echo intensity to magnetic resonance imaging as a metric for tongue fat evaluation. Sleep, 45(2), zsab295. https://doi.org/10.1093/sleep/zsab295